CLINICAL TRIAL: NCT04059822
Title: Effects of Slow and Deep Breathing on Reducing Obstetric Intervention in Women With Pregnancy-induced Hypertension:A Feasibility Study
Brief Title: Slow and Deep Breathing to Lower Blood Pressure in Women With Pregnancy-induced Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding and recruitment
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 251062
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy-Induced Hypertension
Keywords: Slow and deep breathing; Feasibility study
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: All participants will take part in the slow and deep breathing daily exercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Slow and deep breathing (Experimental): Daily practice of slow and deep breathing for 10 minutes per day. Breathing frequency will be 6 breaths per minute, with participants accessing a video aid to help guide their breathing. Breathing exercises will be conducted from enrolment until birth (maximum ~20 weeks if enrolment at 20 weeks gestation until ~40 weeks gestation birth)
  Interventions: Other: Slow and deep breathing

INTERVENTIONS:
Other: Slow and deep breathing — Please see arm description

SUMMARY:
This study evaluates the effect of slow and deep breathing on lowering blood pressure in women with pregnancy-induced hypertension. Slow and deep breathing will be practised daily for 10 minutes from enrolment until the woman gives birth. This feasibility study aims to investigate the practicality of conducting a proposed future randomised controlled trial.

DETAILED DESCRIPTION:
In addition to the slow and deep breathing intervention the women will undertake a short protocol investigating the physiological responses to slow and deep breathing during their initial meeting. The women will undertake 4 separate 5-min breathing exercises with a 5 minute rest period between each exercise. The breathing exercises are normal breathing, and fixed breathing frequencies of 4, 6 and 8 breaths per minute. Blood pressure, heart rate and breathing rate will be monitored continuously, and non-invasively, throughout each breathing protocol.

The women will also have the opportunity to provide feedback on the intervention and their experiences in an online survey at 36 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pregnancy-induced hypertension (PIH). Defined as "new hypertension presenting after 20 weeks of pregnancy without significant proteinuria (urinary protein:creatinine ratio greater than 30mg/mmol" by NICE guidelines (2010) OR diagnosed as having one-off high blood pressure but at risk of developing PIH;
* Single pregnancy;
* Capable of giving informed consent;
* Age over 18.

Exclusion Criteria:

* Under 18 years old;
* Referred immediately to obstetric-care after PIH diagnosis for an immediate intervention, with systolic blood pressure over 160 mmHg or diastolic blood pressure over 100 mmHg;
* Multiple pregnancy (twins, triplets, etc.);
* Current smoker;
* Current diagnosis of respiratory diseases; asthma, COPD (Chronic Obstructive Pulmonary disease), bronchitis. (A previous occurrence or diagnosis that has not been present for longer than 1 year ago does not exclude participants, i.e. childhood asthma);
* Allergy/reaction to gel used on ECG tabs;
* Vulnerable participants who are unable to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Adherence to the breathing exercise intervention | Up to 22 weeks (From enrolment to giving birth)
  Proportion of days breathing exercise completed per participant and average proportion of days breathing exercise completed

SECONDARY OUTCOMES:
Proportion of women referred to obstetric-led care | Up to 22 weeks (From enrolment to giving birth)
  Referral to obstetric-led care will be on the grounds of a test result of 30 mg/mmol^1 in a spot urinary protein, symptom exacerbation and/or increase in systolic and/or diastolic blood pressure

OTHER OUTCOMES:
Proportion of women eligible to participate in study | 5 months (From start to end of recruitment period)
  Proportion of women eligible to participate in the study (using inclusion and exclusion criteria) against number of women who attend the antenatal unit for high blood pressure
Recruitment rates of participation using a hospital antenatal unit | 5 months (From start to end of recruitment period)
  Proportion of women participating in the study against number of eligible women who attend the antenatal unit
Proportion of women who would be willing to be randomised in future trials | Between gestational age 36 weeks and birth. If participant gives birth prior to 36 weeks they will be invited to participate in the questionnaire when appropriate, but before 36 weeks
  Proportion of women who would be willing to be randomised in a future trial (asked in post-questionnaire) against those who would not be willing to be randomised
Adherence to self-monitoring of daily blood pressure | Up to 22 weeks (From enrolment to giving birth)
  Proportion of days blood pressure recorded per participant and average proportion of days blood pressure recorded
Proportion of women withdrawing | Up to 22 weeks (From enrolment to giving birth)
  Proportion of women who do not contribute data due to premature delivery, drop-out or worsening high blood pressure
Difference in blood pressure | Up to 22 weeks (From enrolment to giving birth)
  Average week 1 blood pressure compared with average last week blood pressure (last week prior to giving birth)
Practicality of protocol in delivering slow and deep breathing as an intervention to treat high blood pressure during pregnancy. | Between gestational age 36 weeks and birth. If participant gives birth prior to 36 weeks they will be invited to participate in the questionnaire when appropriate, but before 36 weeks
  Women's perceptions of the intervention, as assessed using the post-questionnaire. The questionnaire includes open ended questions on experiences and barriers to completing the intervention. Likert scale (strongly agree, agree, uncertain, disagree, strongly disagree) questions are also included.
Heart rate responses to slow and deep breathing | Day 1
  Differences in heart rate between breathing protocols (5 minutes of breathing at 4, 6, and 8 breaths per minute and normal breathing)
Blood pressure responses to slow and deep breathing | Day 1
  Differences in blood pressure between breathing protocols (5 minutes of breathing at 4, 6, and 8 breaths per minute and normal breathing)
Stroke volume responses to slow and deep breathing | Day 1
  Differences in stroke volume between breathing protocols (5 minutes of breathing at 4, 6, and 8 breaths per minute and normal breathing)
Cardiac output responses to slow and deep breathing | Day 1
  Differences in cardiac output between breathing protocols (5 minutes of breathing at 4, 6, and 8 breaths per minute and normal breathing)

CONTACTS AND LOCATIONS:
Overall Officials: Malika Felton, Principal Investigator — Postgraduate Researcher
Locations (2):
- United Kingdom (2):
  - Bournemouth University, Bournemouth
  - University Hospitals Dorset NHS Foundation Trust, Poole

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felton M, Hundley VA, Grigsby S, McConnell AK. Effects of slow and deep breathing on reducing obstetric intervention in women with pregnancy-induced hypertension: a feasibility study protocol. Hypertens Pregnancy. 2021 Feb;40(1):81-87. doi: 10.1080/10641955.2020.1869250. Epub 2021 Jan 19. PMID 33463384